CLINICAL TRIAL: NCT07184372
Title: Radiofrequency 448khz in Patients Post Covid 19 With Respiratory Sequelae.
Brief Title: Radiofrequency in Patients Post Covid 19 With Respiratory Sequelae.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Gema Leon (Other)
Responsible Party: Principal Investigator, GEMA LEÓN BRAVO, Gema León Bravo, Clinica Gema Leon
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ART-GLB-RF-RESP-COVID
Record Dates: First submitted 2025-09-17; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: COVID-19; Respiratory Disease; Dyspnea; Cough
Keywords: dyspnea; post covid 19; radiofrequency 448khz; respiratory sequelae; cough
MeSH Terms: conditions — COVID-19; Respiration Disorders; Dyspnea; Cough

STUDY DESIGN:
Intervention Model Description: Longitudinal and experimental
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): The radiofrequency is turn off during the treatment
  Interventions: Other: Placebo
- Conventional Group (Active Comparator): Manual tecniques are applied to improve lung capacity
  Interventions: Other: Manual tecniques
- Experimental Group (Experimental): Manual tecniques and radiofrequency are applied to improve lung capacity
  Interventions: Other: Radiofrequency and manual tecniques

INTERVENTIONS:
Other: Radiofrequency and manual tecniques — We apply manual tecniques while we use the radiofrequency, the treatment is divided into 3 phases:
  * PHASE 1: With the patient in the supine position, treatment was performed along the diaphragm for 10 minutes, of which 5 minutes were spent with the capacitive electrode and the other 5 minutes with the resistive electrode. The plate was placed on the back at the level of the diaphragm.
  * PHASE 2: The patient was placed in the lateral decubitus position on their right side and 3 minutes were spent with the capacitive electrode and 7 minutes with the resistive electrode. The patient was asked to breathe costal-diaphragmatically throughout the entire duration of the resistive electrode. The plate was placed on the right side, at lung level.
  * PHASE 3: The same procedure was performed as in the second phase, only this time on the contralateral side, i.e., on the left side.
  Arms: Experimental Group
Other: Manual tecniques — Manual techniques are used to increase inspiratory capacity, working on the diaphragm and rib cage to increase their mobility along with breathing exercises.
  Arms: Conventional Group
Other: Placebo — The radiofrequency is turn off
  Arms: Placebo group

SUMMARY:
The sequelae that occur in post-COVID-19 patients are multiple and, at a therapeutic level, these represent a new challenge within the general context of the pandemic that the world is suffering.

The virus has managed to end thousands of lives today and many other cases are being charged as directly responsible for a multiplicity of multisystem damages that need to be diagnosed and treated. Among the most relevant, are those that can affect to respiratory levels in patients without previous pahologies, and in patients at risk who already had a pathology prior to infection.

On the other hand, signs and symptoms have been observed characteristic in the organ systems described above in post-contagion patients, directly associated with sequelae SARV-CoV2. The radiofrequency (RF) of electromagnetic waves represents a technology of proven efficacy and safety in multiple fields of both human and veterinary medicine.

These include neurological pathologies, respiratory disease and very especially those that affect the locomotor system. In therapeutics there are different RF modalities depending on the modality, polarity, type of signal and frequency, which in turn translate into different therapeutic profiles, clinical indications, efficacy and safety.

Among the RF technologies most used today and that have a greater scientific background, is the one known as Resistive Capacitive Monopolar RadioFrequency at 448 kHz (INDIBA®) (RFMCR). This study aims to assess the efficacy and safety of RFMCR in the treatment of respiratory sequelae in patients presenting this type of pathologies that appear after contagion by COVID-19. Through this non-invasive technique, the investigators want to show that RF can help the physical rehabilitation of these patients through metabolic stimulation, increased vascularization and oxygenation of directly affected tissues, effects of deep hyperthermia generated by the interaction of the current with the treated biological substrate, as well as the activationof tissue regeneration, the result of subthermal action. It is thus intended to improve signs such as lung capacity, dyspnea, neuropathies and global muscle capacity, which are essential for the recovery of the post-COVID-19 patients.

The hypothesis of this study is that current post-COVID-19 treatments can be significantly improved in order to prevent complications and ensure the patients' well-being.

DETAILED DESCRIPTION:
The new post-pandemic era has left sequelae in patients who presented the signs and symptoms of SARS-CoV-2 and subsequently faced a positive for COVID-19. Such sequelae will be evident at various systemic levels of the affected patienta in the short, medium and long term future. One of these levels is respiratory complications and injuries that have been documented throughout all scientific research since the beginning of passive infections worldwide.

SARS-CoV-2 is transmitted by penetrating the respiratory route (mostly), by fluid contact, and to a lesser extent, through the ocular pathway. In the field of neurology system, different forms of RF, nerve infiltrations, lymph node injuries, plantar fasciitis, spinal (peripheral) nerve disorders, etc. have been documented.

If the investigators focus on one of the most prevalent symptoms (those that affect the respiratory system), the bibliography that endorses that the RFMCR could improve has been referenced.

The aim of this study is to evaluate the efficacy of combined manual therapy and 448 kHz radiofrequency treatment in the recovery of lung capacity in patients with post-COVID-19 sequelae. The work proposed here aims to demonstrate the advantages of establishing RF as an excellent treatment for post-COVID-19 sequelae, due to its ability to reinforce immune action, modulate the inflammatory response and activate cellular and tissue regeneration.

The specific objectives of this research work are:

1. To analyze the evolution of lung capacity using an espirometry in patients treated with the combined protocol.

2. To evaluate the improvement in dysnea and tough 3. To determine the impact of treatment on quality of life. 4. To examine the tolerance, safety and possible side effects of the combined treatment in post-COVID-19 patients. REGULATIONS

1. This clinical study will be carried out in accordance with the protocol, the principles established in the current revised version of the Declaration of Helsinki (Fortaleza, 2013) and in accordance with the applicable regulatory requirements.
2. The researcher is aware, when signing the protocol, of the obligation to adhere to the instructions and procedures described in it, and will ensure that the established provisions are strictly adhered to.
3. The study will not begin until the approval of the Research Ethics Committee has been obtained.
4. The principal investigator is responsible for ensuring that this protocol, the informed consent document, and any other information that is presented or facilitated to the possible subjects is reviewed and approved by the CEI. The Researcher agrees to allow direct access to the REC to all relevant documents.

   INFORMED CONSENT.
5. In this case, patients must give their consent prior to being included in the study. The content and the procedure for obtaining it must be in accordance with all applicable legal requirements.
6. The investigator is responsible for obtaining the written informed consent of each patient participating in this study, after having explained in an understandable way, the nature, objectives, methods, expected benefits and possible risks of the study. The investigator must also explain to them that patients are completely free to refuse to participate in the study or to withdraw from it at any time, for whatever reason.
7. The study patients will give their consent, signing the corresponding model. For this purpose, each informed consent must be signed by both the investigator and the patient.

   CONFIDENTIALITY.
8. All information related to the study is considered confidential in compliance with the confidentiality and custody of the data collected, in accordance with the 3/2018 Law on the protection of personal data (LOPDGDD), (article 5). Article 5.1 .f) of the RGPD states that personal data will be treated in such a way as to guarantee confidentiality and integrity
9. In order to guarantee the confidentiality of the study data, only the main researcher and her team of collaborators will have access to it, the CEI and the pertinent health authorities.

FINANCING

1. The financing is assumed by the Gema León Physiotherapy and Rehabilitation Clinic. There is no direct economic consideration for this, although there is a dedication of time and work by the team of physiotherapists (social security, payroll, personal income tax, etc.) that is not economically remunerated and is assumed or absorbed this way. In addition, the RFMCR technology (equipment and accessories) will be provided by the company INDIBA S.A., through a temporary assignment without any financial compensation either from the Gema León Physiotherapy Clinic, or from any patient. The treatment of these is completely free for them.
2. The patient must travel to the clinic facilities and it is the researcher who will be responsible for the treatment in it.
3. No difficulties are foreseen in its performance since it will be carried out using a schedule adapted to the patient that allows the study to be monitored.

It is intended to carry out a longitudinal study with the participation of 96 patients with lung capacity alterations, who confirmed a positive test for COVID-19. The sample size for our study is large enough to detect a clinically important difference in the primary outcome (s). For this, the investigators reviewed references at the bibliographic level, in which paired studies obtained a statistically significant value, being able to support our study.

If the sample size was insufficient but statistically significant, the investigators would resort to expanding the sample.

The participants were divided into three groups:

* Group 1 or Placebo: the radiofrequency is turn off during the treatment
* Group 2 or conventional: Respiratory manual tecniques are carried out during the treatments to improve lung capacity
* Group 3 or experimental: Radiofrequency 448kz and manual tecniques are applied. They will be evaluated at the beginning, a second evaluation after 3 weeks and a third final control after 12 sessions. A fourth evaluation will be carried out after the last and final evaluation, 6 weeks after finishing the treatment.

Each of the participants will be informed of the study, the objective, its possible benefits and the side effects that could arise. A) Therefore, each patient must give their free and confirmed consent through signature. Among the items in the methodology, the following stand out:

Primary outcome: Spirometry was performed at the beginning of the first, sixth, and twelfth sessions, and one and a half months after completing treatment. All spirometry tests were performed in the same manner: the patient was seated with their feet flat on the floor and a nose clip was placed on the patient and they were asked to take two normal breaths, and on the third, to take a maximum inhalation and a maximum exhalation. We obteined the following parameters: FVC (Forced Vital Capacity), FEV1 (Forced Expiratory Volume in 1 Second), FVC/FEV1 (Ratio of FVC to volume expired in 1 second), PEF (Peak Expiratory Flow), PEFT (Peak Expiratory Flow Time), FEF50% (Forced expiratory flow at 50% of expiration), FEF25% - FEF75% (Forced expiratory flow between 25% and 75% of expiration), FEF50%/FIF50 (Ratio of forced expiratory flow at 50% of expiration to forced inspiratory flow at 50% of inspiration) and FEV1/FEV0.5 (Ratio of forced expiratory volume in 1 second to forced expiratory volume in the first 0.5 s)

Secondary outcome: The Sadoul Dyspnea Scale is internationally validated to evaluate the feeling of the patient´sdyspnea and has a 6-grade classification: Grade 0 (No dyspnea), Grade 1 (Dyspnea after significant exertion or climbing two flights of stairs), Grade 2 (Dyspnea when climbing one flight of stairs or with brisk walking on a slight incline), Grade 3 (Dyspnea during brisk walking on level ground), Grade 4 (Dyspnea occurs with slow walking), Grade 5 (Dyspnea with minimal exertion)

Tertiary outcome: Chest measuremnets. All chest measurements, were taken at the first and last measurement sessions, following the same protocol. These measurements were taken with the subject standing in a neutral position and at three different levels, using the following reference points at each level: the axillary line, the tip of the xiphoid bone, and the level of the tenth rib. In addition, three measurements were taken at each level at maximum inspiration, maximum expiration, and neutral.

The therapeutic protocol will be executed in the facilities of the Gema León Physiotherapy and Rehabilitation Clinic (Cordoba, Spain). Depending on the group of treatments the protocol will consist in:

* Group 1 or Placebo: the radiofrequency is turn off during the treatment
* Group 2 or conventional: Respiratory manual tecniques are carried out during the treatments to improve lung capacity,
* Group 3 or experimental: the same manual tecniques of the group 2 are applied while we use the radiofrequency. We divide the treatment in 3 phases:

PHASE 1: With the patient in the supine position, treatment was performed along the diaphragm for 10 minutes, of which 5 minutes were spent with the capacitive electrode and the other 5 minutes with the resistive electrode. The plate was placed on the back at the level of the diaphragm.

PHASE 2: The patient was placed in the lateral decubitus position on their right side and 3 minutes were spent with the capacitive electrode and 7 minutes with the resistive electrode. The patient was asked to breathe costal-diaphragmatically throughout the entire duration of the resistive electrode. The plate was placed on the right side, at lung level.

PHASE 3: The same procedure was performed as in the second phase, only this time on the contralateral side.

Such RF therapeutic protocol will be implemented by application with an INDIBA® Activ device, whose function is to reduce inflammation, stimulate immunity and promote tissue regeneration. This will consist of a 45-minute treatment. A total of 12 sessions will be scheduled (two per week), and all processes will be documented from the beginning of therapy (the resources used will be provided by INDIBA and the Gema León Physiotherapy and Rehabilitation Clinic, whose supervision will be carried out by the direction of both).

Another variables which they are gonna be take into account are sex, age, weight, height, smoker, vaccination, number of days with symptoms and type of symptom.

The statistical analysis is based on variables of nominal type mostly, which are suitable for the Chi square test with a significance value of 95% for the results (p <0.05). However, if there are numerical data that must be compared between groups, the analysis will be used for ANOVA test with the same significance value for the comparison between results.

ELIGIBILITY:
Inclusion Criteria:

* have passed covid 19
* have respiratory sequelae after covid 19 during more than a month
* have dyspnea, cough or fatigue

Exclusion Criteria:

* be pregnant
* have pacemaker
* have or had passes thrombosis
* have a respiratory disease before covid

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Spirometry | 3 months
  spirometry tests were performed in the same manner: the patient was seated with their feet flat on the floor and a nose clip was placed on the patient and they were asked to take two normal breaths, and on the third, to take a maximum inhalation and a maximum exhalation. We obteined the following parameters: FVC (Forced Vital Capacity), FEV1 (Forced Expiratory Volume in 1 Second), FVC/FEV1 (Ratio of FVC to volume expired in 1 second), PEF (Peak Expiratory Flow), PEFT (Peak Expiratory Flow Time), FEF50% (Forced expiratory flow at 50% of expiration), FEF25% - FEF75% (Forced expiratory flow between 25% and 75% of expiration), FEF50%/FIF50 (Ratio of forced expiratory flow at 50% of expiration to forced inspiratory flow at 50% of inspiration) and FEV1/FEV0.5 (Ratio of forced expiratory volume in 1 second to forced expiratory volume in the first 0.5 s

SECONDARY OUTCOMES:
Sadoul Dyspnea Scale | 3 months
  The Sadoul Dyspnea Scale is internationally validated to evaluate the feeling of the patient´sdyspnea and has a 6-grade classification: Grade 0 (No dyspnea), Grade 1 (Dyspnea after significant exertion or climbing two flights of stairs), Grade 2 (Dyspnea when climbing one flight of stairs or with brisk walking on a slight incline), Grade 3 (Dyspnea during brisk walking on level ground), Grade 4 (Dyspnea occurs with slow walking), Grade 5 (Dyspnea with minimal exertion)
Leiscester Test | 3 months
  It is a questionnaire used to objectively assess chronic cough and its effect on quality of life. It is structured into three domains: physical, psychological, and social.
Chest measurements | 3 months
  All chest measurements, were taken at the first and last measurement sessions, following the same protocol. These measurements were taken with the subject standing in a neutral position and at three different levels, using the following reference points at each level: the axillary line, the tip of the xiphoid bone, and the level of the tenth rib. In addition, three measurements were taken at each level at maximum inspiration, maximum expiration, and neutral.

CONTACTS AND LOCATIONS:
Overall Officials: Gema León Bravo, Fisioterapia, Principal Investigator — Gema León Physiotherapy and Rehabilitation Clinic
Locations (1):
- Clinica de Fisioterapia Gema Leon, Córdoba, Cordoba, Spain

IPD SHARING:
Plan to Share IPD: No
The request for the data will be studied and considered upon prior and justified request